CLINICAL TRIAL: NCT07166211
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of CM512 Injection in Subjects With CSU
Brief Title: Study of CM512 Injection in Subjects With Chronic Spontaneous Urticaria(CSU)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM512-112101
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Spontaneous Urticaria (CSU)
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: CM512 injection
- Group 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: CM512 injection — subcutaneous injection
  Arms: Group 1
Drug: placebo — subcutaneous injection
  Arms: Group 2

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled phase II clinical study to evaluate the efficacy, safety, pharmacokinetics, pharmacodynamics, and immunogenicity of CM512 in subjects with CSU.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the Informed Consent Form.
* Age ≥ 18 years old and ≤ 75 years old.
* Patients with a diagnosis of CSU before screening visit, and the duration was ≥6 months.
* Pruritus and wheals existed for more than 6 weeks before screening, despite regular H1-Antihistamines(AH) treatment during this period.
* A stable dose of the second-generation H1-Antihistamines(AH) has been continuously used for at least 3 days before screening, and the individual is willing to continue to use it stably as stipulated in the protocol during the study period.
* Within 7 days before randomization, UAS7≥16 and ISS7 ≥8.

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Planned major surgical procedure during the patient's participation in this study.
* Has ever experienced a systemic allergic reaction or immediate allergic reaction to any biological product (including any excipients).
* CM512 has been used before.
* Women who are pregnant or breastfeeding. During the study period, subjects who had plans to have children, or did not agree to contraception.
* With any medical or non-medical conditions that are not suitable for participation in this study by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-11-02 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline in 7-day urticaria activity score (UAS7) at 16 weeks of treatment (W16) | Up to 16 weeks
  UAS7 is a verified and recognized Patient Reported Outcomes(PRO) scale for evaluating the activity of CSU, consisting of 7-day hives-severity score and 7-day itch-severity score (ISS7), ranging from 0 to 42 points. UAS7 score < 7 indicates low urticaria activity, UAS7 score > 28 suggests high urticaria activity and severe condition.

CONTACTS AND LOCATIONS:
Overall Officials: Litao Zhang, Principal Investigator — Tianjin Academy of Traditional Chinese Medicine Affiliate Hospital; Zuotao Zhao, Study Chair — Tianjin Academy of Traditional Chinese Medicine Affiliate Hospital
Locations (1):
- Tianjin Academy of Traditional Chinese Medicine Affiliate Hospital, Tianjin, Tianjin Municipality, China